CLINICAL TRIAL: NCT07085676
Title: A Phase 1 Dose Escalation and Safety Study of HBI0101 CART in B-cell Mediated Refractory Autoimmune Diseases
Brief Title: Phase 1 Study of HBI0101 CAR-T in Refractory B-Cell Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Polina Stepensky (Other)
Responsible Party: Sponsor-Investigator, Polina Stepensky, Prof. Polina Stepensky, Director Department of Bone Marrow Transplantation and Cancer Immunotherapy, Hadassah Medical Organization, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI0101 ARD 001
Record Dates: First submitted 2025-05-06; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus (SLE); Systemic Sclerosis (SSc); Idiopathic Inflammatory Myopathy (IIM); Rheumatoid Arthritis (RA)
Keywords: B-cell mediated autoimmune rheumatic diseases; Systemic Lupus Erythematosus (SLE); Systemic sclerosis (SSC); Idiopathic inflammatory myopathy (IIM); Rheumatoid arthritis (RA); B-cell maturation antigen (BCMA); Autologous CAR-T
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Myositis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CART (Experimental): Each subject subjects will receive a single dose of 450 x 10^6 or 800 x 10^6 BCMA CART cells
  Interventions: Biological: HBI0101 CART

INTERVENTIONS:
Biological: HBI0101 CART — HBI0101 CART is defined as autologous T cells transduced ex-vivo with anti-BCMA CAR retroviral vector encoding the chimeric antigen receptor (CAR) targeted to human BCMA. The HBI0101 CART may be provided fresh or cryopreserved.

SUMMARY:
A Phase 1 study of HBI0101 BCMA-CART in B-Cell Mediated Autoimmune Rheumatic Diseases. The goal of the study is evaluation of safety and identification of the maximum HBI0101 CART dose that may be administered safely to patients with B-cell mediated autoimmune disease.

DETAILED DESCRIPTION:
Up to 60 subjects with B-cell mediated autoimmune rheumatic diseases will be enrolled in a single-arm, open-label, single-site Phase 1 study.

The study includes 2 parts. The first Part A is an establishment of the safety profile followed by a dose ranging, maximum tolerated dose (MTD) study and the second Part B is an extension phase to further evaluate safety at the selected safe dose.

Eligible subjects will undergo leukapheresis procedure to provide starting material for manufacturing of HBI0101 CART investigational product. Each eligible subject will receive a single dose of HBI0101 CART cells. Prior to administration of HBI0101 CART, the study subjects will undergo lymphodepletion. Following administration of HBI0101 CART the subjects will be hospitalized for several days and then will return for routine follow-up periodical visits until 48 months after infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~65 years old
2. Diagnosis of B-cell mediated autoimmune rheumatic diseases - SLE, SSc, IIM, RA.
3. Expected survival period ≥ 3 months;
4. Serum creatinine <221.0μmol/L (2.5mg/dl);
5. AST/ALT below 3 times the upper limit of normal, blood bilirubin <34.2 μmol/L (2.0 mg/dl);
6. Cardiopulmonary function is basically normal, echocardiography indicates that the ejection fraction is >45%, normal to mild pulmonary hypertension, and the oxygen saturation is above 93% in the resting state without oxygen;
7. No obvious active infection;
8. Physical fitness score 0~2 points (ECOG standard);
9. There are suitable veins for blood cell apheresis or whole blood collection, and there are no contraindications for blood collection;
10. Women of childbearing age should have a negative serum or urine pregnancy test 48 hours before CAR T cell reinfusion, and agree to take effective contraceptive measures during the trial until the last follow-up;
11. Voluntary participation and informed consent signed by the patient or his/her legal/authorized representative;

Exclusion Criteria:

1. CNS disease-currently active severe CNS, including cerebritis, cerebrovascular accident (CVA), and seizures.
2. Kidney disease-hemodialysis, Serum creatinine >221.0μmol/L (2.5mg/dl);
3. Abnormal liver function: aspartate transaminase (AST) or alanine transaminase (ALT) or glutamyl transpeptidase (GGT) detection value is greater than 3 times the upper limit of normal (ULN); or alkaline phosphatase (ALP) or total bilirubin test value greater than 1.5 times the upper limit of normal (ULN); Exceptional: liver function disturbance due to myositis
4. Cardiovascular disease: Unstable angina or myocardial infarction or coronary artery bypass graft (CABG) within 6 months prior to leukapheresis/ moderate- severe pulmonary hypertension/ severe arrhythmia (ventricular tachycardia, ventricular fibrillation, high grade ventricular block) in the past 6 months; New York heart function class (NYHA) class III- Level IV or LVEF<45%.
5. Lung disease: patients with interstitial lung disease (ILD) with any of the following: *Requiring O2 therapy and or FVC≤45% of predicted or DLCO≤40% of predicted at screening. * Evidence of pulmonary hypertension as defined as estimated RVSP> 50 mmHg.
6. Muscle disease: evidence of any of the following: * Severe proximal muscle atrophy of upper or lower extremity on MRI or clinical examination. *Finding of muscular inflammation or myopathy other than the indication, such as inclusion body myositis (IBM), or cancer-associated myositis (myositis diagnosed within 2 years of cancer).
7. Other uncontrolled diseases: acute diseases (such as acute pneumonia or other infection, pulmonary embolism, diabetic ketoacidosis, acute pancreatitis, etc.) that are clinically unstable or have not been effectively controlled and are not related to SLE/SSc/IIM/RA which in the judgment of the investigator may confound study results or place subjects at undue risk.
8. Biologics therapy: Received biologic therapy (antibody, inhibitor or agonist) targeting T, B lymphocytes, cytokines or receptors within two months before the study or Rituximab therapy within six months before the study.
9. Participated in any clinical study within 3 months prior to enrollment, or participate in other clinical investigations during the study period.
10. Received live vaccine treatment within 30 days prior to Visit 2;
11. Previous or concurrent malignancy with the following exceptions: Adequately treated basal cell or squamous cell carcinoma, in situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to screening. A primary malignancy which has been completely resected, or treated, and is in complete remission for at least 5 years prior to screening.
12. Transplantation: History of vital organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/or bone marrow transplantation.
13. HIV positive.
14. Active hepatitis B or C.
15. Pregnant or lactating women.
16. Inability to understand or follow the research protocol subject requirements.
17. Have any other clinically significant disease history or current disease that, in the judgment of the research physician, may pose a risk to the safety of the subjects, or interfere with the completion of the research procedure and the evaluation of safety and efficacy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) | 21 days after infusion
  MTD will be determined by dose limiting toxicities, defined as any HBI0101 CART-related Grade 3 to 5 toxicity occurring after infusion of the investigational product.
Confirmation of safety with selected dose (at or below MTD) | 21 days after infusion
  MTD will be determined by dose limiting toxicities, defined as any HBI0101 CART-related Grade 3 to 5 toxicity occurring after infusion of the investigational product

SECONDARY OUTCOMES:
Overall survival | 3 months for up to 24 months, every 6 months for up to 48 months
  Evaluation of overall survival
Four-year progression free survival: All Cohorts | 4 years following infusion
  Survival without evidence of relapse or disease progression
Disease-specific response/progression endpoints: Systemic Lupus Erythematosus (SLE) cohort | 4 years following infusion
  Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) < 4 (no disease activity)
Disease-specific response/progression endpoints: Systemic Lupus Erythematosus (SLE) cohort | 4 years following infusion
  Serologic response: presence of positive ANA, anti-dsDNA and anticardiolipin antibody titers
Disease-specific response/progression endpoints: Systemic Lupus Erythematosus (SLE) cohort | 4 years following infusion
  Serologic response: abnormal complement C3 and C4 levels
Disease-specific response/progression endpoints: Systemic Scleroderma (SSc) cohort | 4 years following infusion
  Skin condition: An improvement is indicated by a decrease on modified Rodan Skin Score (mRSS) of ≥ 5 points
Disease-specific response/progression endpoints: Systemic Scleroderma (SSc) cohort | 4 years following infusion
  Pulmonary function: Change in forced vital capacity (FVC), total lung capacity (TLC) or diffusing capacity of the lung for carbon monoxide (DLCO) > 10%
Disease-specific response/progression endpoints: Idiopathic Inflammatory Myopathies (IIM) cohort | 4 years following infusion
  Myositis disease activity assessment visual analogue scale (MDAAT) score >5% absolute change in core set measures
Disease-specific response/progression endpoints: Idiopathic Inflammatory Myopathies (IIM) cohort | 4 years following infusion
  Muscle condition: Manual Muscle test >5% absolute change in core set measures
Disease-specific response/progression endpoints: Idiopathic Inflammatory Myopathies (IIM) cohort | 4 years following infusion
  Disease related biomarker: Creatine Kinase (CPK)
Disease-specific response/progression endpoints: Rheumatoid Arthritis (RA) cohort | 4 years following infusion
  RA-reaching low disease activity (DAS28CRP) ≤2.7
Disease-specific response/progression endpoints: Rheumatoid Arthritis (RA) cohort | 4 years following infusion
  Serologic response: RF (rheumatoid factor) and/or ACPA (anti-citrullinated protein antibody) positivity

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah MO, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kfir-Erenfeld S, Asherie N, Grisariu S, Avni B, Zimran E, Assayag M, Sharon TD, Pick M, Lebel E, Shaulov A, Cohen YC, Avivi I, Cohen CJ, Stepensky P, Gatt ME. Feasibility of a Novel Academic BCMA-CART (HBI0101) for the Treatment of Relapsed and Refractory AL Amyloidosis. Clin Cancer Res. 2022 Dec 1;28(23):5156-5166. doi: 10.1158/1078-0432.CCR-22-0637. PMID 36107221
- [Background] Asherie N, Kfir-Erenfeld S, Avni B, Assayag M, Dubnikov T, Zalcman N, Lebel E, Zimran E, Shaulov A, Pick M, Cohen Y, Avivi I, Cohen C, Gatt ME, Grisariu S, Stepensky P. Development and manufacture of novel locally produced anti-BCMA CAR T cells for the treatment of relapsed/refractory multiple myeloma: results from a phase I clinical trial. Haematologica. 2023 Jul 1;108(7):1827-1839. doi: 10.3324/haematol.2022.281628. PMID 36200421